CLINICAL TRIAL: NCT01930994
Title: A Pharmacokinetic Study to Compare Sino-implant (II) During Four Years of Use to Jadelle During Five Years of Use by Kenyan Women
Brief Title: Kenya Sino-implant (II) PK Study
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient numbers of Sino-implant users available for study participation.
Sponsor: FHI 360 (Other)
Collaborators: Marie Stopes International (Other)
Responsible Party: Sponsor
Other Study IDs: 475139
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Contraception
Keywords: LNG: Levonorgestrel; MSI: Marie Stopes International; MSK: Marie Stopes Kenya; PK: Pharmacokinetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Cohort 1: Twenty Sino-implant (II) and twenty Jadelle users enrolled 1-3 months before their 6-month insertion anniversary.
- Cohort 2: TwentySino-implant (II) and twenty Jadelle users enrolled 1-3 months before their 12-month insertion anniversary;
- Cohort 3: Twenty Sino-implant (II) and twenty Jadelle) users enrolled 1-3 months before their 24-month insertion anniversary
- Cohort 4: Twenty Sino-implant(II) and twenty Jadelle users enrolled 1-3 months before their 36-month insertion anniversary;
- Cohort 5: Forty Sino-implant (II) and forty Jadelle users enrolled 1-3 months before their 48-month insertion anniversary;
- Cohort 6: Forty Jadelle users enrolled 2-6 months before their 60-month insertion anniversary.

SUMMARY:
A cross-sectional study to compare pharmacokinetics of Sino-implant (II) during four years of used and Jadelle during five years of use by Kenyan women.

DETAILED DESCRIPTION:
A cross-sectional study to compare the pharmacokinetics of Sino-implant (II) during four years of use and Jadelle during five years of use by Kenyan women. The active ingredient in both implants is levonorgestrel (LNG) which is a synthetic progestin that has been used in combined oral contraceptives and in progestin-only pills for more than 30 years.

Population: A total of 280 women between the ages of 18 to 44 years who are currently using Sino-implant (II) or Jadelle contraceptive implants will be enrolled in one of six cohorts of women:

Cohort 1: (n=20 Sino-implant (II), n=20 Jadelle) women enrolled 1-3 months before their 6-month insertion anniversary.

Cohort 2: (n=20 Sino-implant (II), n=20 Jadelle) women enrolled 1-3 months before their 12-month insertion anniversary.

Cohort 3: (n=20 Sino-implant (II), n=20 Jadelle) women enrolled 1-3 months before their 24-month insertion anniversary.

Cohort 4: (n=20 Sino-implant (II), n=20 Jadelle) women enrolled 1-3 months before their 36-month insertion anniversary.

Cohort 5: (n=40 Sino-implant (II), n=40 Jadelle) women enrolled 1-3 months before their 48-month insertion anniversary.

Cohort 6: (n=40 Jadelle) women enrolled 2-6 months before their 60-month insertion anniversary.

Women in all cohorts will be followed for up to 6 months.

Study Duration: Up to 6 months of participant recruitment and up to 6 months elapsed after the baseline visit for the second study visits. 15 months total in the field including training, study initiation, recruitment, follow-up, and close-out.

Two blood samples spaced 2 to 6 months apart will be drawn from each woman for hormone measurements.

Primary Objective: To compare total and free levonorgestrel (LNG) plasma concentrations at four years of Sino-implant (II) use to total and free LNG plasma concentrations at five years of Jadelle use in Kenyan women

Secondary Objectives:

1. To compare total and free LNG plasma concentrations at four years of Sino-implant (II) use to total and free LNG plasma concentrations at four years of Jadelle use
2. To characterize the total and free LNG plasma concentration-time profiles over four years following Sino-implant (II) and over five years following Jadelle insertion
3. To characterize the sex hormone binding globulin (SHBG) serum concentration-time profile over four years following Sino-implant (II) and over five years following Jadelle insertion

ELIGIBILITY:
Inclusion Criteria:

* Have a Sino-implant (II) or Jadelle implant set in place, confirmed by physical exam;
* Have a confirmed contraceptive implant insertion date consistent with the criteria for the cohort she is to be enrolled in;
* Be aged between 18 and 44 years, inclusive;
* Not wish to become pregnant in the next six months;
* Not desire implant removal within the next six months.
* Be able to understand the information given to them and to make personal decisions on whether to participate or not in the study;
* Consent to participation, and sign an informed consent form;
* Agree and be able to return to the clinic for the second study visit.

Exclusion Criteria: The following criteria exclude participation in the study:

* Use of rifampicin, and/or anticonvulsants (barbiturates, phenytoin, phenobarbital, carbamazepine, oxcarbazepine, primidone, topiramate), and/or herbal products containing St. John's wort (Hypericum perforatum), by self-report;7
* Use of medications containing LNG or other hormones that impact LNG or SHBG disposition, e.g. treatment with LNG or oral contraceptives for bleeding disturbances, by self-report;
* Use of anti-retroviral drugs, by self-report;
* Any condition (social or medical) which in the opinion of the Investigator would make study participation unsafe, would interfere with adherence to study requirements or complicate data interpretation.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 18 and 44 who have received contraceptive implants from the Marie Stopes Kenya Eastleigh clinic and MSK mobile clinics in the Nairobi area.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Total and Free LNG concentrations in Jadelle users at Four Years and Sino-implant users at Five Years | 6 months
  Total and free LNG plasma concentrations measured at four years of Sino-implant (II)use and at five years of Jadelle use

SECONDARY OUTCOMES:
Total and Free LNG concentrations at Four Years of Jadelle and Sino-implant Use | 6 months
  Total and free LNG plasma concentrations at 4 years of Sino-implant (II) use and total and free LNG plasma concentrations at 4 years of Jadelle use
Total and free LNG plasma concentration-time profiles at 4 years following Sino-implant (II) and at over 5 years following Jadelle insertion | 6 months
  Total and free LNG plasma concentration-time profiles at 4 years of Sino-implant(II)use compared to over 5 years of Jadelle use
SHBG serum concentration-time profile over 4 years following Sino-implant (II) and over 5 years following Jadelle insertion. | 6 months
  SHBG serum concentration-time profile at at 4 years of Sino-implant(II)use compared to over 5 years of Jadelle use

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ayallo, MD, Principal Investigator — Marie Stopes Kenya
Locations (1):
- Marie Stopes Kenya Eastleigh Clinic, Nairobi, Kenya